CLINICAL TRIAL: NCT01013038
Title: Thrombus Aspiration During Percutaneous Coronary Intervention in Acute Non-ST-elevation Myocardial Infarction Study (TAPAS II)
Brief Title: Thrombus Aspiration During Percutaneous Coronary Intervention in Acute Non-ST-elevation Myocardial Infarction Study
Acronym: TAPAS II
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Netherlands Heart Foundation (Other)
Responsible Party: Marthe Anna Kampinga, MD & Felix Zijlstra, MD PhD, University Medical Center Groningen, Thoraxcenter
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008B101
Record Dates: First submitted 2009-11-06; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Non-ST-Elevation Myocardial Infarction
Keywords: myocardial infarction; percutaneous coronary intervention; thrombus aspiration
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional percutaneous coronary intervention (Active Comparator)
  Interventions: Procedure: conventional PCI
- Thrombus aspiration (Experimental)
  Interventions: Procedure: Thrombus aspiration followed by stent implantation

INTERVENTIONS:
Procedure: Thrombus aspiration followed by stent implantation — Export aspiration catheter 6F (Medtronics)
  Arms: Thrombus aspiration
Procedure: conventional PCI — balloon angioplasty and/or stent implantation
  Arms: Conventional percutaneous coronary intervention

SUMMARY:
In this trial, the investigators will evaluate the effect of thrombus aspiration followed by stent implantation in improving myocardial blush grade in patients with acute non-ST-elevation myocardial infarction compared to conventional percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
The Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS) has shown that thrombus aspiration improves myocardial perfusion and clinical outcome compared to conventional primary percutaneous coronary intervention (PCI) in patients with ST-segment elevation myocardial infarction. Impaired myocardial perfusion due to spontaneous or angioplasty-induced embolization of atherothrombotic material also occurs in patients with Non-ST-elevation myocardial infarction (NSTEMI). The aim of this study is to determine whether thrombus aspiration before stent implantation will result in improved myocardial perfusion in patients with NSTEMI compared to conventional PCI.

The study is a single-centre, prospective, randomised trial with blinded evaluation of endpoints. The planned inclusion is 540 patients with acute NSTEMI who are candidates for urgent PCI.

If thrombus aspiration leads to significant improvement of myocardial perfusion in patients with acute NSTEMI it may become part of the standard interventional approach.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute NSTEMI defined by

  * Chest pain suggestive for myocardial ischemia for at least 30 minutes,
  * Time from onset of symptoms of less than 72 hours
  * ECG with ST-segment shifts (depression of >0.1 mV in at least two contiguous leads or transient ST-segment elevation >0.1 mV in at least two contiguous leads for less than 30 minutes) and/or T-wave changes (inversion of >0.15 mV in at least two contiguous leads)
  * Positive cardiac troponin T >0,01 μg/L.
* Clinical indication for urgent PCI of the ischemia-related target lesion as identified at coronary angiography

Exclusion Criteria:

* Persistent ST-elevation of more than 0.1 mV in 2 or more leads
* Presence of cardiogenic shock
* Inability to obtain informed consent
* Known existence of a life-threatening disease with a life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2007-12; Primary Completion 2011-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of myocardial blush grade 3 after PCI | During PCI procedure

SECONDARY OUTCOMES:
Coronary angiographic outcomes | During PCI procedure
Histopathological outcomes of atherothrombotic material | After inclusion is stopped: mean 1 year (storage at -80 degrees Celcius)
Enzymatic infarct size | During hospital stay
Electrocardiographic outcomes | 30 to 60 minutes after PCI
Clinical outcomes at 30 days and 1 year | 30 days till 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands